CLINICAL TRIAL: NCT00070629
Title: Promune™ (CPG 7909 Injection) In Combination With Chemotherapy In Patients With Advanced Or Metastatic Non-Small Cell Lung Cancer, A Randomized, Multi-Center, Controlled, Phase 2 Study
Brief Title: CPG 7909 Injection in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C017; ProMune; CO17; A8501017
Record Dates: First submitted 2003-10-06; First posted 2003-10-08 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: Immunotherapy; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — ProMune; Drug Therapy; Paclitaxel; Docetaxel; Cisplatin; Carboplatin

ARMS (2):
- 1 (Experimental): Chemotherapy (a taxane and a platinum compound) plus CPG 7909 Injection
  Interventions: Drug: CPG 7909; Drug: Chemotherapy
- 2 (Active Comparator): Chemotherapy (a taxane and a platinum compound)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: CPG 7909 — CPG 7909 Injection will be administered subcutaneously at a starting dose of 0.20 mg/kg at the beginning of Weeks 2 and 3 of the three-week cycle.
  Other Names: ProMune, PF-3512676
  Arms: 1
Drug: Chemotherapy — A taxane and a platinum compound given on week one of three-week cycles:
  Regimen A: Paclitaxel 175 mg/m2 over 1 - 3 hrs, Cisplatin 75 mg/m2 Regimen B: Paclitaxel 175 mg/m2 over 1 - 3 hrs, Carboplatin AUC of 6 Regimen C: Docetaxel 75 mg/m2, Cisplatin 75 mg/m2 Regimen D: Docetaxel 75 mg/m2, Carboplatin AUC of 6
  Arms: 2
Drug: Chemotherapy — A taxane and a platinum compound given on week one of three-week cycles:
  Regimen A: Paclitaxel 175 mg/m2 over 1 - 3 hrs, Cisplatin 75 mg/m2 Regimen B: Paclitaxel 175 mg/m2 over 1 - 3 hrs, Carboplatin AUC of 6 Regimen C: Docetaxel 75 mg/m2, Cisplatin 75 mg/m2 Regimen D: Docetaxel 75 mg/m2, Carboplatin AUC of 6
  Other Names: Paclitaxel (Taxol), docetaxel (TAXOTERE) cisplatin and carboplatin (e.g. PARAPLATIN)
  Arms: 1

SUMMARY:
Eligible patients will be randomized in a ratio of 2:1 to receive either chemotherapy (a taxane and a platinum compound) plus CPG 7909 Injection or chemotherapy alone. Protocol therapy will be administered until disease progression or intolerable toxicity. CpG 7909 Injection will be administered subcutaneously, on Weeks 2 and 3 of each three-week cycle (days 8 and 15) and chemotherapy will be administered on Week 1 (Day 1). Patients will undergo complete disease evaluation at the end of every other treatment cycle until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer that is beyond surgical cure or that is metastatic (Stage IIIB or IV according to AJCC).
* Patients must have measurable disease according to the RECIST criteria.

Exclusion Criteria:

* Prior treatment with chemotherapy; patients may have received prior radiotherapy.
* Patients with suspected or known CNS metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2003-05; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Efficacy- overall response rate (CR & PR) according to the RECIST criteria | Indeterminate
Safety- drug exposure, adverse events, laboratory tests, vital signs, ECG, and physical examinations | Indeterminate

SECONDARY OUTCOMES:
Secondary Efficacy | Indeterminate
compare number of patients who achieve complete response, partial response, or stable disease (CR, PR, SD) between the two treatment groups | Indeterminate
duration of overall response (CR, PR), survival time, and time to disease progression. | Indeterminate
To assess the immunopharmacodynamic response to CPG 7909 Injection plus chemotherapy in responding vs nonresponding patients receiving chemotherapy or the combination. | Indeterminate

CONTACTS AND LOCATIONS:
Locations (24):
- United States (17):
  - Office of Ronald Yanagihara, Gilroy, California
  - Kenmar Research Institute, LLC, Los Angeles, California
  - Comprehensive Cancer Center of the Dessert, Palm Springs, California
  - Florida Cancer Specialist, Fort Myers, Florida
  - Indiana Hematology and Oncology Associates, Indianapolis, Indiana
  - Medical Center Vincennes, Vincennes, Indiana
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - Southeast Nebraska Hematology Oncology Consultants, PC, Lincoln, Nebraska
  - VA New Jersey Health Care System, East Orange, New Jersey
  - HemOnCare, Brooklyn, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - Cancer Care Institute of Carolina, Aiken, South Carolina
  - Charleston Hematology/Oncology, PA, Charleston, South Carolina
  - The Family Cancer Center, Collierville, Tennessee
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (3):
  - Queen Elizabeth II Health, Halifax, Nova Scotia
  - Ottawa Regional Cancer Center, Ottawa, Ontario
  - McGill University, Montreal, Quebec
- Germany (4):
  - Staedtisches Krankenhaus Martha-Maria, Halle-Dolau
  - Universitätsklinikum Mannheim der Universität Heidelberg, Heidelberg
  - St. Vincentius-Kliniken gAG, Hamatologie-Onkologie, Karlsruhe
  - Klinikum Rechts der Isar, München